CLINICAL TRIAL: NCT04451226
Title: A Single-Arm Phase 3 Clinical Study to Investigate the Long-Term Safety of Fezolinetant in Women in China Suffering From Vasomotor Symptoms (Hot Flashes) Associated With Menopause
Brief Title: A Study to Assess the Safety and Tolerability of Fezolinetant in Women Seeking Treatment for Relief of Vasomotor Symptoms (VMS) Associated With Menopause
Acronym: Moonlight 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2693-CL-0307; CTR20200676 (Registry Identifier: ChinaDrugTrials.org.cn)
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Hot Flashes
Keywords: Vasomotor Symptoms; menopause; fezolinetant; ESN364
MeSH Terms: conditions — Hot Flashes | interventions — fezolinetant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fezolinetant (Experimental): Participants will receive fezolinetant 30 milligrams (mg) orally once daily for 52 weeks.
  Interventions: Drug: Fezolinetant

INTERVENTIONS:
Drug: Fezolinetant — Oral
  Other Names: ESN364; VEOZAH

SUMMARY:
This study is for women in menopause with hot flashes. Menopause, a normal part of aging, is the time of a woman's last period. Hot flashes can interrupt a woman's daily life. The purpose of this study is to find out how safe it is for these women to take fezolinetant long term (up to 52 weeks). To do that, the study will look at the number and severity of the "adverse events." Those are the side effects that study participants have while they are in the study. The study treatment is fezolinetant (1 tablet of fezolinetant) once a day. The study participants will take study treatment for 52 weeks. At weeks 2 and 4 and then once a month, the study participants will go the hospital or clinic for a check-up. They will be asked about medications, side effects and how they feel. Other checks will include physical exam and vital signs (heart rate, temperature and blood pressure). Blood and urine will be collected for laboratory tests. At some study visits, study participants will complete questionnaires that are about their quality of life. Study participants who still have their uterus will have 2 more tests done at the first and last study visits. One of the 2 tests is endometrial biopsy. This test involves removing a small amount of tissue from the inside lining of the uterus. The tissue is then checked under a microscope. The other test is transvaginal ultrasound. It uses sound waves to create pictures of the organs in the pelvis. The sound waves are transmitted by a probe (transducer), which is placed inside the vagina. Study participants may have a screening mammogram done at the first and/or last study visit. A mammogram is an x-ray picture of the breasts used to screen for breast cancer. Study participants who did not have this test done in the last 12 months will have it done at the first study visit. They will have it done at the last study visit if they are due for their screening mammogram and their own doctor agrees. The last check-up at the hospital or clinic will be 3 weeks after the last dose of study treatment.

DETAILED DESCRIPTION:
The study will consist of a screening period, a 52-week treatment period and a follow-up visit, 3 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index ≥ 16 kg/m^2 and ≤ 38 kg/m^2 at the screening visit.
* Subject confirmed as menopausal per 1 of the following criteria at the screening visit:

O Subject has spontaneous amenorrhea for >= 12 consecutive months O Spontaneous amenorrhea for ≥ 6 months with biochemical criteria of menopause (follicle-stimulating hormone [FSH] > 40 International Units per Liter [IU/L], or O Having had bilateral oophorectomy ≥ 6 weeks prior to the screening visit (with or without hysterectomy).

O FSH > 40 IU/L if subjects received hysterectomy but still have ovary

* Subject is seeking treatment for relief for VMS associated with menopause.
* Subject is in good general health as determined on the basis of medical history and general physical examination, including a bimanual clinical pelvic examination and clinical breast examination devoid of relevant clinical findings, performed at the screening visit; hematology and biochemistry parameters; pulse rate and/or blood pressure; and ECG within the reference range for the population studied, or showing no clinically relevant deviations.
* Subject has documentation of a normal/negative or no clinically significant abnormal findings on mammogram (or echo) (e.g., <BI-RADS class 4; obtained at screening or within the prior 12 months of screening). Appropriate documentation includes a written report or an electronic report indicating normal/negative or no clinically significant abnormal findings.
* Subject is willing to undergo a transvaginal ultrasound (TVU) to evaluate the uterus and ovaries at screening and at week 52 (end of treatment). For subjects who are withdrawn from the study prior to completion, a TVU should be collected at the early discontinuation (ED) visit. This is not required for subjects who have had a partial (supra-cervical) or full hysterectomy.
* Subject is willing to undergo an endometrial biopsy at screening and at week 52 (end of treatment) or the ED visit if endometrial thickness > 4 millimeter (mm) indicated by TVU; and subject is willing to undergo an endometrial biopsy at any time during the study in the case of uterine bleeding. This is not required for subjects who have had a partial (supra-cervical) or full hysterectomy. A biopsy with insufficient material for evaluation, or unevaluable material, is acceptable provided the endometrial thickness is no greater than 8 mm.
* Subject has documentation of a normal or not clinically significant abnormal Papanicolaou (Pap) test (or equivalent cervical cytology) within the previous 12 months of screening or at screening. This is not required for subjects who have had a full hysterectomy.
* Subject has a negative urine pregnancy test at screening.
* Subject has a negative serology panel (including hepatitis B virus surface antigen [HBs] and hepatitis C virus antibody [anti-HCV], and human immunodeficiency virus [HIV]) at screening.
* Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject uses a prohibited therapy (strong and moderate cytochrome P450 [CYP] 1A2 inhibitors, hormone replacement therapy [HRT], hormonal contraceptive, any treatment for VMS [prescription, over the counter or herbal]) or is not willing to wash out and discontinue such drugs for the full extent of the study.
* Subject has a known substance abuse or alcohol addiction within 6 months of screening.
* Subject has a history of a malignant tumor, except for non-metastatic basal cell carcinoma of the skin.
* Subject has uncontrolled hypertension, defined as systolic blood pressure >= 140 millimeters of mercury (mmHg) or diastolic blood pressure as >= 90 mmHg based on an average of 2 to 3 readings within the screening period.

O Subjects with a medical history of hypertension who are well controlled may be enrolled.

O Subjects who do not meet the criteria may, be re-assessed after initiation or review of antihypertensive measures.

* Subject has a history of severe allergy, hypersensitivity, or intolerance to drugs in general, including the study drug and any of its excipients.
* For subjects with a uterus: Subject has an unacceptable result from the TVU assessment at screening, i.e., full length of endometrial cavity cannot be visualized or presence of a clinically significant abnormal finding.
* For subjects with an endometrial thickness > 4 mm as indicated by TVU at screening: Subject has an endometrial biopsy confirming presence of disordered proliferative endometrium, endometrial hyperplasia, endometrial cancer, or other clinically significant abnormal findings in the at screening. A biopsy with insufficient material for evaluation, or unevaluable material is acceptable provided the endometrial thickness is no greater than 8 mm.
* Subject has a history of an undiagnosed uterine bleeding within the last 6 months of screening.
* Subject has a history of seizures or other convulsive disorders.
* Subject has a medical condition or chronic disease (including history of neurological [including cognitive], hepatic, renal, cardiovascular, gastrointestinal, pulmonary [e.g., moderate asthma], endocrine, or gynecological disease) or malignancy that could confound interpretation of the study outcome.
* Subject has active liver disease, jaundice, or elevated liver aminotransferases (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]), elevated total or direct bilirubin, elevated international normalized ratio (INR), or elevated alkaline phosphatase (ALP) at screening. Subject with mildly elevated ALT or AST up to 1.5 × the upper limit of normal (ULN) can be enrolled if total and direct bilirubin are normal. Subject with mildly elevated ALP (up to 1.5 × ULN) can be enrolled if cholestatic liver disease is excluded and no cause other than fatty liver is diagnosed. Subject with Gilbert's syndrome with elevated total bilirubin (TBL) may be enrolled as long as hemolysis is ruled out (i.e., direct bilirubin (DBL), hemoglobin and reticulocytes are normal).
* Subject has creatinine > 1.5 × ULN; or estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease formula <= 59 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2) at the screening visit.
* Subject has a history of suicide attempt or suicidal behavior within the prior to 12 months of study enrollment or has suicidal ideation within the prior to 12 months of study enrollment (a response of "yes" to questions 4 or 5 on the suicidal ideation portion of the C-SSRS), or who is at significant risk to commit suicide at screening and at visit 2.
* Subject has previously been enrolled in a clinical trial with fezolinetant.
* Subject has received an investigational study drug within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subject is unable or unwilling to complete the study procedures.
* Subject has any condition which, makes the subject unsuitable for study participation.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Up to 55 weeks
  An adverse event (AE) is any untoward medical occurrence in a participant administered a study drug, and which does not necessarily have to have a causal relationship with this treatment.
Number of Participants With Adverse Events Based on Severity | Up to 55 weeks
  An AE is any untoward medical occurrence in a participant administered a study drug, and which does not necessarily have to have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Change From Baseline in Endometrial Thickness | Baseline and 52 weeks
  Endometrial thickness is a measure of how thick the lining of the uterus is. Change from baseline will be reported.
Percentage of Participants With Endometrial Hyperplasia and/or Endometrial Cancer | Up to 52 weeks
  Endometrial hyperplasia is thickening of the lining of the uterus. Endometrial cancer is cancer of the lining of the uterus. Percentage of participants will be reported.
Number of Participants With Vital Sign Abnormalities and/or Adverse Events (AEs) | Up to 55 weeks
  Number of participants with potentially clinically significant vital sign values.
Number of Participants With Laboratory Value Abnormalities and/or Adverse Events (AEs) | Up to 55 weeks
  Number of participants with potentially clinically significant laboratory values.
Number of Participants With Suicidal Ideation and/or Behavior as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to 55 weeks
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinician administered assessment tool that evaluates suicidal ideation and behavior. Number of participants that have an affirmative response provided to the 5 items for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods (not plan) without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and/or to the 5 items for suicidal behavior (1. Preparatory acts or behavior, 2. Aborted attempt, 3. Interrupted attempt, 4. Actual attempt, 5. Completed suicide) will be reported.
Number of Participants With Electrocardiogram (ECG) Abnormalities and/or Adverse Events (AEs) | Up to 52 weeks
  Number of participants with potentially clinically significant ECG values.
Change From Baseline in Bone Specific Alkaline Phosphatase (BSAP) Levels | Baseline, week 52 and week 55
  Change from baseline in serum concentrations of BSAP will be reported.
Change From Baseline in Procollagen Type 1 Amino-terminal Propeptide (P1NP) Levels | Baseline, week 52 and week 55
  Change from baseline in serum concentrations of P1NP will be reported.
Change From Baseline in Carboxy-terminal Telopeptide of Type I Collagen (CTX) Levels | Baseline, week 52 and week 55
  Change from baseline in serum concentrations of CTX will be reported.
Change From Baseline in Serum Concentration of Sex Hormones | Baseline, week 4, week 12, week 24 , week 52 and week 55
  Change from baseline in serum concentration of sex hormones will be reported.
Change From Baseline in Sex Hormone-Binding Globulin (SHBG) | Baseline, week 4, week 12, week 24 , week 52 and week 55
  Change from baseline in serum concentration of SHBG will be reported.
Pharmacokinetics (PK) of Fezolinetant in Plasma: Concentration | Week 4, week 12, week 24 and week 52
  Concentration will be recorded from the PK plasma samples collected.
Pharmacokinetics (PK) of Fezolinetant Metabolite ES259564 in Plasma: Concentration | Week 4, week 12, week 24 and week 52
  Concentration will be recorded from the PK plasma samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma China, Inc.
Locations (29):
- China (29):
  - Site CN86002, Beijing
  - Site CN86015, Beijing
  - Site CN86029, Beijing
  - Site CN86032, Chengdu
  - Site CN86001, Guangzhou
  - Site CN86019, Guangzhou
  - Site CN86022, Guangzhou
  - Site CN86040, Guangzhou
  - Site CN86042, Guangzhou
  - Site CN86008, Hangzhou
  - Site CN86012, Hangzhou
  - Site CN86005, Hunan
  - Site CN86039, Jiangsu
  - Site CN86010, Jinlin
  - Site CN86020, Kunming
  - Site CN86037, Liuchow
  - Site CN86006, Nanjing
  - Site CN86007, Nanjing
  - Site CN86018, Nanning
  - Site CN86034, Ningxia Hui Nationality Autonomous Region
  - Site CN86009, Shanghai
  - Site CN86011, Shanxi
  - Site CN86004, Shenzhen
  - Site CN86028, Shijiazhuang
  - Site CN86026, Suzhou
  - Site CN86038, Taiyuan
  - Site CN86030, Tianjin
  - Site CN86036, Tianjin
  - Site CN86025, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as compounds terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Yu Q, Ming F, Ma J, Cai Y, Wang L, Ren M, Zhang J, Ma X, Miyazaki K, He W, Wang X. Long-term safety of fezolinetant in Chinese women with vasomotor symptoms associated with menopause: the phase 3 open-label MOONLIGHT 3 clinical trial. J Int Med Res. 2024 May;52(5):3000605241246624. doi: 10.1177/03000605241246624. PMID 38818887
- See also: Link Description: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14545&tenant=MT_AST_9011